CLINICAL TRIAL: NCT04417413
Title: Safety and Efficacy of Non-ablative Er:YAG Laser Therapy for the Treatment of Pelvic Organ Prolapse and Coexisting Stress Urinary Incontinence: A Retrospective Case Series.
Status: Completed | Type: Observational
Sponsor: Aleksandra Novakov Mikic (Other)
Responsible Party: Sponsor-Investigator, Aleksandra Novakov Mikic, Prof Dr, Poliklinika Novakov i saradnici
Organization: Poliklinika Novakov i saradnici (Other)
Other Study IDs: POP+SUI
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cystocele; Pelvic Organ Prolapse; Stress Urinary Incontinence
MeSH Terms: conditions — Cystocele; Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fotona ProlapLase — Non-ablative SMOOTH mode intravaginal Er:YAG teratment for pelvic organ prolapse

SUMMARY:
The objective of the study is to retrospectively collect the data on patients who underwent pelvic organ prolapse treatment using a non-ablative Er:YAG laser with SMOOTH mode and to conduct an objective evaluation of safety and efficacy of Er:YAG laser treatment. In a group of patients that have concomitant stress urinary incontinence symptoms, the effectiveness of the treatments on these symptoms will be evaluated as well.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) and stress urinary incontinence (SUI) affect many women and can dramatically decrease their quality of life. Most of the patients diagnosed with stress urinary incontinence also have a degree of pelvic organ prolapse and vice-versa.

One of the more promising new approaches in treating disorders connected to pelvic floor dysfunction has been the introduction of vaginal erbium laser treatment for pelvic organ prolapse.

The primary aim of the present retrospective study was toassess the effectiveness of vaginal erbium laser with SMOOTH mode for the treatment of patients with pelvic organ prolapse and co-existing stress urinary incontinence, if present.

ELIGIBILITY:
Inclusion Criteria:

All patients that had pelvic organ prolapse with or without concomitant stress urinary incontinence and that were treated using non-ablative Fotona Er:YAG laser (ProlapLase treatment) in the time period from 2015 to 2016 will be included in this retrospective study.

Exclusion Criteria:

Patients who failed to attend a follow-up appointment will be excluded from this retrospective case series study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that had pelvic organ prolapse with or without concomitant stress urinary incontinence and that were treated using non-ablative Fotona Er:YAG laser (ProlapLase treatment) in the time period from 2015 to 2016 were included in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Cystocele stage | Before and at all follow ups (up to 3 months after last treatment)
  Assesment of POP grade using Baden-Walker scale
Severity of stress urinary incontinence | Before and at all follow ups (up to 3 months after last treatment)
  assessment of SUI severity using ICIQ-UI questionnaire

SECONDARY OUTCOMES:
Assesment of safety | Before and at all follow ups (up to 3 months after last treatment)
  Assesment of adverse effects
Patient satisfaction | Before and at all follow ups (up to 3 months after last treatment)
  Assesment of patient satisfaction using 0-10 VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinika Novakov i sar., Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No